CLINICAL TRIAL: NCT07361692
Title: Study of the Effectiveness of Transcranial Direct Current Stimulation (tDCS) in the Management of Complex Regional Pain Syndrome
Brief Title: Effectiveness of Transcranial Direct Current Stimulation (tDCS) in the Management of Complex Regional Pain Syndrome
Acronym: ALGOSTIM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Polyclinique de l'Europe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-20-ESN
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Complex Regional Pain Syndrome (CRPS)
Keywords: Transcranial direct current stimulation; Complex Regional Pain Syndrome; pain; quality of life; anxiety; central sensitization
MeSH Terms: conditions — Complex Regional Pain Syndromes; Pain; Anxiety Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient group receiving tDCS stimulation (Experimental): Progressive increase in stimulation intensity up to 2 mA, then continuation at a plateau for a total of 20 minutes, then a decrease in stimulation intensity for 30 seconds at the end of the session before an automatic stop.
  Interventions: Other: transcranial direct current stimulation
- Patient group receiving tDCS placebo stimulation (Placebo Comparator): Control group : The stimulation intensity is gradually increased up to 2 mA for 1 minute, then decreased to zero stimulation. A further increase in stimulation is programmed 10 minutes after the start of stimulation.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: transcranial direct current stimulation — progressive increase in stimulation intensity up to 2 mA, then continuation at a plateau for a total of 20 minutes, then a decrease in stimulation intensity for 30 seconds at the end of the session before an automatic stop.
  Arms: Patient group receiving tDCS stimulation
Other: Placebo — The stimulation intensity is gradually increased up to 2 mA for 1 minute, then decreased to zero stimulation. A further increase in stimulation is programmed 10 minutes after the start of stimulation.
  Arms: Patient group receiving tDCS placebo stimulation

SUMMARY:
Transcranial direct current stimulation (tDCS) is a non-invasive therapy increasingly used in facilities treating patients with chronic pain. This complementary therapy has the advantage of being non-pharmacological, with transient and mild side effects, an excellent safety profile, and good efficacy in the contexts where it has been the subject of dedicated research: neuropathic pain, fibromyalgia, and visceral pain. Few studies have focused on the application of tDCS in the context of complex regional pain syndrome (CRPS), which is a common condition.

DETAILED DESCRIPTION:
This protocol aims to compare a group receiving a tDCS protocol with a sham control group. The hypothesis of this study is that tDCS is effective in treating CRPS in terms of reducing pain and the functional and emotional consequences of pain.

The primary objective of the study is to evaluate the effectiveness of tDCS on pain in patients with CRPS (complex regional pain syndrome), measured by the numerical pain scale (EN), after one month of treatment and one month after the end of treatment, compared to the sham arm.

The secondary objectives are:

* To assess anxiety and depression symptoms (HAD)
* To assess the functional impact of pain (Concise Pain Questionnaire - QCD)
* To assess central sensitization (Central Sensitization Inventory - CSI)
* To identify adverse effects related to tDCS

ELIGIBILITY:
Inclusion Criteria:

* Major
* Clinically active or active complex regional pain syndrome (CRPS) with positive Budapest criteria
* Scintigraphy showing signs consistent with CRPS
* Being affiliated with or a beneficiary of a social security scheme

Exclusion Criteria:

* Algodystrophy no longer meeting the Budapest criteria
* Relative contraindication to tDCS: psychosis (including treated psychosis), uncontrolled epilepsy, large scalp scar, intracerebral/intracranial metallic body
* Pregnant or breastfeeding women
* Minors
* Persons under legal protection (guardianship, conservatorship, and protective supervision)
* Persons deprived of their liberty by judicial or administrative order
* Unwilling individuals who cannot give their consent or cannot return for scheduled visits according to the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Analog Visual Scale | one month post treatment